CLINICAL TRIAL: NCT02636907
Title: Assessment of Real-life Patient Handling Experience of BI 695501 Administered Subcutaneously With an Autoinjector in Patients With Rheumatoid Arthritis: an Open-label, Interventional Clinical Trial Followed by an Extension Phase of BI 695501 Administered With a Prefilled Syringe
Brief Title: Assessment of the Handling Experience With the BI 695501 Autoinjector in Patients With Rheumatoid Arthritis Followed by an Extension Phase Using BI 695501 Prefilled Syringe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1297.11; 2015-003030-27 (EudraCT Number)
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

ARMS (1):
- BI 695501 (Experimental)
  Interventions: Drug: BI 695501 Autoinjector; Drug: BI 695501 Prefilled syringe

INTERVENTIONS:
Drug: BI 695501 Autoinjector
Drug: BI 695501 Prefilled syringe

SUMMARY:
This is an open-label, phase II study of BI 695501 to assess handling experience of patients with Rheumatoid Arthritis using an autoinjector. The extension phase is to provide patients with additional exposure to BI 695501 and to enhance the safety database for this compound.

ELIGIBILITY:
Inclusion criteria:

* Moderately to severely active Rheumatoid arthritis (RA) for at least 6 months, which is not adequately controlled by non-biologics DMARDs.
* No contraindications to anti-Tumor necrosis factor (TNF) agents.
* Either biologics naive or biologics-experienced but with no experience of self-administration medication using autoinjector or pen.
* Patients must be able and willing to self-inject BI 695501. Further inclusion criteria apply.

Exclusion criteria:

* Experience with self-administration of medication using an autoinjector or pen.
* American College of Rheumatology functional Class IV or wheelchair/ bed bound.
* Primary or secondary immunodeficiency.
* History of tuberculosis (TB). Further exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2016-06-21 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (19):
- United States (9):
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Lovelace Scientific Resources, Incorporated, Venice, Florida
  - Klein and Associates, M.D., P.A., Cumberland, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - Metroplex Clinical Research Center, Dallas, Texas
  - Rheumatology Clinic Of Houston, P.A., Houston, Texas
  - Arthritis & Osteoporosis Associates LLP, Lubbock, Texas
  - Heartland Research Associates, LLC, Nassau Bay, Texas
- Poland (10):
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Wojewodzki Szpital Zespolony w Elblagu, Elblag
  - Medica Pro Familia Spolka Akcyjna, Oddzial w Gdyni, Gdynia
  - Medical Centre Pratia Katowice I, Katowice
  - Medical Centre Pratia Krakow, Krakow
  - Specialist Center ALL-MED, Krakow, Krakow
  - Niepubliczny ZOZ, "Nasz Lekarz", Lekarzy Rodzinnych z, Torun
  - Medical Centre Pratia Warszawa, Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw

REFERENCES:
- [Derived] Cohen S, Klimiuk PA, Krahnke T, Assudani D. Successful administration of BI 695501, an adalimumab biosimilar, using an autoinjector (AI): results from a Phase II open-label clinical study (VOLTAIRE(R)-RL). Expert Opin Drug Deliv. 2018 Jun;15(6):545-548. doi: 10.1080/17425247.2018.1472572. Epub 2018 May 15. PMID 29764238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An Open-label, Interventional clinical trial followed by an extension phase of BI 695501 in patients with Rheumatoid Arthritis.
  EoT: End of treatment (EoT)
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be entered to trial drug if any of the specific entry criteria was violated.
Groups:
- BI 695501: Patients were administered BI 695501 solution for injection (40 milligram (mg)/0.8 milliliter (mL)) by subcutaneous injection every 2 weeks using an autoinjector (7-week Autoinjector Assessment Period) or Prefilled syringe (PFS) (optional 42-week Extension Phase). Patients were treated with up to 26 injections.
Period: Autoinjector Assessment Period
Arm/Group | BI 695501
Started | 77 (Assigned to treatment.)
Completed | 73 (Completed autoinjector assessment period (Day 50).)
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Period: Extension Phase
Arm/Group | BI 695501
Started | 72
Completed | 62
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF): The SAF contained all patients in the all subjects enrolled set (ENR) who received at least 1 dose of trial drug or attempted to inject it as indicated by the questionnaire on self-injection with autoinjector.
Arm/Group | BI 695501
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.4 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Autoinjector Assessment Period: Percentage of Successful Self-injections as Reported in the Questionnaires Completed by Both the Trial Site Personnel and the Patient Analysing All Self-injections
Description: The percentage of successful self-injections as reported in the questionnaires completed by both the trial site personnel and the patient during the Autoinjector Assessment Period analyzing all self-injections occurring after the training self-injection up to the EoT Visit. Successful self-injections were based on the response to Question 2 (Q2) on the questionnaire, which queried whether the full content of the autoinjector was injected into the body. An injection was considered successful when both the patient and the qualified trial site personnel responded yes to the Q2 on their respective questionnaires. If they responded no to Q2, patients and trial site personnel were instructed to also answer Question 3, which asked what prevented the patient for injecting the full contents of the autoinjector. Planned injections after discontinuation from the trial were not included in the analysis.
  Percentage of injections calculated relative to the total number of first injections.
Time Frame: Up to Day 50.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of injections
Arm/Group | BI 695501
Number analyzed (Participants) | 77
Percentage of injections | 99.1 [96.72 to 99.75]

2. Secondary Outcome: Autoinjector Assessment Period: Percentage of Any Autoinjector Handling Events
Description: The percentage of any autoinjector handling event during the self-injection process included any one of the following events which prevented the patient from successfully self-injecting the full content of the autoinjector and which occurred after the training self-injection up to the EoT Visit: removing the cap of the autoinjector (3a); pressing the injection button of the autoinjector (3b); or holding the autoinjector down against the skin until the injection is completed (3c).
  Percentage of injections was calculated relative to the total number of injections (both unsuccessful and successful).
Time Frame: Up to Day 50.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of injections
Arm/Group | BI 695501
Number analyzed (Participants) | 77
Percentage of injections
  Unsuccessful | 0.9
  Successful | 99.1

3. Secondary Outcome: Autoinjector Assessment Period: The Percentage of Patients With Local Injection Site Reactions
Description: Qualified trial site personnel contacted the patient 48 hours after each self-injection during the autoinjector assessment period to collect all Adverse Events (AEs), including injection-site reactions. Data is reported as Treatment-Emergent AEs (TEAEs), defined as AEs that started or worsened on or after the first dose of trial medication during the treatment period and prior to the last date of trial medication during treatment period + 10 weeks (70 days) inclusive. The autoinjector assessment period started on the first autoinjector administration date (Day 1 visit) and ended on Day 50 visit date (included). If a TEAE occurred in the 10 weeks after the last autoinjector administration but prior to the first injection during the extension phase, it was to be accounted for in the autoinjector assessment period.
  Percentage of subjects calculated relative to the total number of subjects in the analysis set.
Time Frame: Up to 17 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501
Number analyzed (Participants) | 77
Percentage of participants | 6.5

4. Secondary Outcome: Autoinjector Assessment Period: The Percentage of Patients With Drug-related Adverse Events Per Investigator Assessment
Description: A treatment-related TEAE was defined as any TEAE assessed by the investigator as related to the trial medication. Data is reported for the autoinjector assessment period. TEAEs were defined as AEs that started or worsened on or after the first dose of trial medication during the treatment period and prior to the last date of trial medication during treatment period + 10 weeks (70 days) inclusive. The autoinjector assessment period started on the first autoinjector administration date (Day 1 visit) and ended on Day 50 visit date (included). If a TEAE occurred in the 10 weeks after the last autoinjector administration but prior to the first injection during the extension phase, it was to be accounted for in the autoinjector assessment period.
Time Frame: Up to 17 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501
Number analyzed (Participants) | 77
Percentage of participants | 11.7

5. Secondary Outcome: Autoinjector Assessment Period and Extension Phase: The Percentage of Patients With Local Injection Site Reactions
Description: The percentage of patients with local injection site reactions in the Autoinjector assessment period and Extension Phase. In Extension phase, patients were given diaries to record events between each site visit during extension phase. Patients were instructed to accurately record the following on the diary cards: the dates & times of BI 695501 dosing; problems encountered with dosing; the occurrence of any AEs; the use of concomitant therapies; and the PFS storage conditions. Patients were instructed to contact the site if they experienced any AEs between designated site visits. In Extension phase Data is reported as Treatment-Emergent AEs (TEAEs), defined as AEs that started or worsened on or after the first PFS administration date (Day 57 visit) and after the 10 weeks of the last dose during the extension phase, it was to be accounted for in the Extension phase treatment period. Percentage of subjects calculated relative to the total number of subjects in the analysis set
Time Frame: up to Week 60
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501
Number analyzed (Participants) | 77
Percentage of participants | 23.4

6. Secondary Outcome: Autoinjector Assessment Period and Extension Phase: The Percentage of Patients With Drug-related Adverse Events as Per Investigator Assessment
Description: The percentage of patients with drug-related adverse events as per investigator in the Autoinjector assessment period and Extension Phase. In Extension phase, Treatment-Emergent AEs (TEAEs), defined as AEs that started or worsened on or after the first dose of trial medication and prior to the last date of trial medication during Extension phase treatment period + 10 weeks (70 days) inclusive. The Extension phase treatment period started on the first PFS administration date (Day 57 visit) and ended on Day 351 visit date (included). Thus If a TEAE occurred from the first PFS administration and after the 10 weeks of the last dose during the extension phase, it was to be accounted for in the Extension phase treatment period.
Time Frame: up to Week 60
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | BI 695501
Number analyzed (Participants) | 77
Percentage of participants | 36.4

ADVERSE EVENTS:
Time Frame: From first drug infusion until 10 weeks after last drug infusion, up to 376 days.
Arm/Group | BI 695501
All-Cause Mortality (participants affected / at risk) | 0/77
Serious Adverse Events (participants affected / at risk) | 9/77
Other Adverse Events (participants affected / at risk) | 40/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 (N=77)
Anaemia (Blood and lymphatic system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Depression (Psychiatric disorders) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Device related infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Drug use disorder (Psychiatric disorders) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Chest pain (General disorders) | 1
Complication associated with device (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 (N=77)
Sinusitis (Infections and infestations) | 6
Headache (Nervous system disorders) | 8
Upper respiratory tract infection (Infections and infestations) | 9
Bronchitis (Infections and infestations) | 5
Viral upper respiratory tract infection (Infections and infestations) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Injection site bruising (General disorders) | 11
Injection site erythema (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.